CLINICAL TRIAL: NCT04352491
Title: An Online Survey to Understand Feelings Related to COVID-19 Among ILBS Patients With Liver Disease (FEELIV COVID)
Brief Title: An Online Survey to Understand Feelings Related to COVID-19 Among ILBS Patients With Liver Disease
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-COVID-03
Record Dates: First submitted 2020-04-14; First posted 2020-04-20 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-04

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with liver disease: All people who have shown at Institute of Liver and Biliary Sciences (1st January 2018 - 31st March 2020), will be sent the SMS for participation.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The current outbreak of COVID-19 pandemic has been marked by severe psychological problems. People around the world experienced a similarly frightening public health emergency, on a global scale, with the spread of this corona infection. (1) Studies of the Severe Acute Respiratory Syndrome (SARS) outbreaks that occurred in Canada, Taiwan, and Hong Kong found that the enormous emotional burden carried by those health care workers who were on the front lines of the battle against the disease led to psychological morbidity like anxiety, stress and even further leads to Post traumatic stress disorder. The initial phase of the COVID-19 outbreak in China in 2020 also reported more than half of the respondents rated the psychological impact as moderate-to-severe, and about one-third reported moderate-to-severe anxiety in general population.(2)

- The chances of Fear, anxiety and stress are even higher in Individuals with preexisting liver disease as they have restriction of services for getting treatment. Moreover, they can have the following additional issues:

* Fear of severe form of Corona present (as presented in most of the media and research)
* Fear of dying
* Added uncertainty
* Family members also worried

DETAILED DESCRIPTION:
* As the Indian Government recommended the public to minimize face-to-face interaction and isolate them at home, potential respondents will be invited through a text message which will lead to a survey monkey page (designed by IT team at ILBS, New Delhi).
* All people who have shown at ILBS (1st January 2018 - 31st March 2020), will be sent the SMS for participation. They will be asked to provide phone numbers for retrieval of their Child-Turcotte-Pugh (CTP) and Model for End Stage Liver Disease (MELD) scores from hospital records. Patients with education more than 10th standard (or able to understand / read English) will only proceed with the survey.
* After clicking the link users will complete an online survey. The first page will give them basic information about the FEELIV-COVID survey and if they consent to participate, they will complete the survey. The decision to undertake the survey voluntarily, and will have no impact on their ongoing treatment.
* Informed consent will be obtained in the form of electronic name entry at the beginning of the survey. Their name entry will be taken as an approval to allow the investigators data regarding their Liver disease. Only the following data will be taken from the patient's records:

  * Child-Turcotte-Pugh (CTP) score
  * Model for End Stage Liver Disease (MELD) score
  * Etiology of Liver Dysfunction
* No other data will be retrieved for the purpose of this study from patient's records.

ELIGIBILITY:
Inclusion Criteria:

- Patients who have shown at Institute of Liver & Biliary Sciences (ILBS) between 1st January 2018 and 31st March 2020 will be considered as currently being enrolled at ILBS for treatment.

Exclusion Criteria:

- Incomplete questionnaires

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have shown at ILBS between 1st January 2018 and 31st March 2020 will be considered as currently being enrolled at ILBS for treatment. Only their data will be used for the purpose of this study.
Sampling Method: Non-Probability Sample
Enrollment: 347 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Assessment of the fear levels during the COVID-19 disease pandemic among patients with Liver disease (currently under treatment from ILBS) | Day 0
  Following questionnaire will be used For Fear of COVID-19: FEAR OF COVID-19 Scale Fear of Coronavirus-19 Scale: The participants indicate their level of agreement with the statements using a five-item Likert-type scale. Answers included "strongly disagree," "disagree," "neither agree nor disagree," "agree," and "strongly agree". The minimum score possible for each question is 1, and the maximum is 5. A total score is calculated by adding up each item score (ranging from 7 to 35). The higher the score, the greater the fear of cororonavirus-19.
Assessment of the anxiety levels during the COVID-19 disease pandemic among patients with Liver disease (currently under treatment from ILBS) | Day 0
  Following questionnaire will be used
  o For, anxiety: DASS - 21 Scale Depression, Anxiety and Stress Scale - 21 Items (DASS-21) Depression Anxiety Stress Scale (DASS)-21: The DASS-21 is based on three subscales of depression, stress, and anxiety and each subscale consists of seven questions each. Each subscale comprises of seven statements regarding how the test subject was feeling over the last week and four responses ranging from 0- did not apply to me at all, 1- applied to me some of the time, 2- applied to me for a considerable amount of time to 3- applied to me very much/most of the time. The scoring system is of the Likert type and the total score for each subscale gives the severity of that very symptom which has a range from 0 to 21 for each subscale.
Assessment of the stress levels during the COVID-19 disease pandemic among patients with Liver disease (currently under treatment from ILBS) | Day 0
  Following questionnaire will be used
  o Stress levels: DASS - 21 Scale Depression Anxiety Stress Asymptomatic ≤4 ≤3 ≤7 Symptomatic >4 >3 >7

SECONDARY OUTCOMES:
Association between presence of Liver disease and fear levels | Day 0
  Following questionnaire will be used
  o For Fear of COVID-19: FEAR OF COVID-19 Scale
Association between presence of Liver disease and anxiety levels | Day 0
  Following questionnaire will be used
  o For, anxiety levels: DASS - 21 Scale Depression, Anxiety and Stress Scale - 21 Items (DASS-21) Higher Scores mean worse condition
Association between presence of Liver disease and stress levels | Day 0
  Following questionnaire will be used
  o For stress levels: DASS - 21 Scale Depression, Anxiety and Stress Scale - 21 Items (DASS-21) Higher Scores mean worse condition.
Correlation between Fear and Child-Turcotte-Pugh Score | Day 0
  Higher Scores mean worse condition
Correlation between anxiety and Child-Turcotte-Pugh Score | Day 0
  Higher Scores mean worse condition
Correlation between stress and Child-Turcotte-Pugh Score | Day 0
  Higher Scores mean worse condition
Correlation between fear and Model for End Stage Liver Disease Score | Day 0
  Higher Scores mean worse condition
Correlation between anxiety and Model for End Stage Liver Disease Score | Day 0
  Higher Scores mean worse condition
Correlation between stress and Model for End Stage Liver Disease Score | Day 0
  Higher Scores mean worse condition

CONTACTS AND LOCATIONS:
Overall Officials: Dr Shiv Kumar Sarin, DM, Study Director — Institute of Liver & Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided